CLINICAL TRIAL: NCT00608985
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Active Reference, Parallel-group Polysomnography Study to Assess the Efficacy and Safety of a 16-day Oral Administration of ACT-078573 in Adult Subjects With Chronic Primary Insomnia
Brief Title: Almorexant (ACT 078573) in Adult Subjects With Chronic Primary Insomnia
Acronym: RESTORA 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Midnight Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-057A301
Record Dates: First submitted 2008-01-11; First posted 2008-02-06 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Primary Insomnia
Keywords: sleeplessness; orexin receptor antagonist; almorexant; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — almorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): almorexant 200 mg
  Interventions: Drug: almorexant
- 2 (Experimental): almorexant 100 mg
  Interventions: Drug: almorexant
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 4 (Active Comparator): zolpidem 10 mg
  Interventions: Drug: zolpidem

INTERVENTIONS:
Drug: almorexant — 2 100 mg almorexant tablets and 1 placebo matching over-encapsulated zolpidem
  Arms: 1
Drug: almorexant — 1 100 mg almorexant tablet, 1 placebo matching almorexant tablet, and 1 placebo matching over-encapsulated zolpidem
  Arms: 2
Drug: Placebo — 2 placebo matching almorexant tablets and 1 placebo matching over-encapsulated zolpidem
  Arms: 3
Drug: zolpidem — 2 placebo matching almorexant tablets and 1 zolpidem 10 mg over-encapsulated
  Arms: 4

SUMMARY:
A polysomnography study to evaluate the effect, safety and tolerability of oral administration of almorexant (ACT 078573) in adult subjects with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-64 years) with a diagnosis of primary insomnia.

Exclusion Criteria:

* History of any sleep disorder, or any Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) axis I disorder other than primary insomnia.
* Sleep apnea, or restless legs syndrome.
* Daytime napping of more than 1 hour per day.
* Important caffeine consumption, heavy tobacco use, alcohol or drug abuse within 2 years prior to the screening visit.
* Unwillingness to refrain from drugs, over-the-counter or herbal medication having an effect on sleep or behavior.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 709 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cluydts, Dr., Study Chair — Cognitive and Biological Psychology, University of Brussels
Locations (91):
- Australia (9):
  - Sleep Disorders Laboratory, Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Adult Sleep Center, Monash Medical Centre, Clayton, Victoria
  - Western Hospitpal, Private Bag, Footscray, Victoria
  - Institute for Breathing and Sleep (IBAS), Heidelburg, Victoria
  - The Woolcock Institute of Medical Research, Glebe
  - Australian Clinical Research Organisation, Kippa-Ring
  - Melbourne Sleep Disorder Centre, Melbourne
  - Burnside Hospital Clinical Trials Centre, Toorak Gardens
  - Westmead Hospital, Department of Respiratory, Westmead
- Austria (3):
  - Medical University of Innsbruck, Department of Neurology, Innsbruck
  - Rudolfinerhaus, Vienna
  - University of Vienna - Department of Neurology, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - CH Jolimont / Sleep Disorders Center, Hospital de Jolimont, Haine-Saint-Paul
  - Clinique Andre Vesale, Montigny Le Tilleuil
- Bulgaria (2):
  - Hospital St. Naum, Paediatr. Neurology, Sofia
  - MHAT 'St. Marina', Varna
- Czechia (5):
  - Oddeleni nasledne pece, Nemocnice Ceske Budejovice, České Budějovice
  - Centrum pro poruchy spanku a bdeni, Neurologicka klinika, Katerinska
  - Fakultni nemocnice Ostrava/Klinika detske neurologie SLEEP LABORATORY, Ostava-Poruba
  - Poradna pro porchy spanku a spankova, Laborator Unimeds s.r.o., Prague
  - Somnocentrum Trutnov-spankova laborator, Oddeleni neurologie, Trutnov
- Denmark (3):
  - Scansleep Aps, Sovnlaegecentret, Aarhus
  - Sovnlagecentret - Scan Sleep, Copenhagen
  - Scan Sleep ApS, Sovnlaegecentret, Copenhagen
- Finland (3):
  - Tutkimuskeskus Vitalmed, Helsinki
  - Unesta Research Center, Tampere
  - University of Turku, Sleep Research Unit, Turku
- France (6):
  - Hopital Pellegrin, Bordeaux
  - Hopital Raymond Poincare, Garches
  - Service de Neurologie B, Hopital Gui de Chauliac, Montpellier
  - Hopital Pitie-Salpetriere, Paris
  - Centre du Sommeil et de la Vigilance, Hopital Hotel Dieu de Paris, Paris
  - Federation des Pathologies du Sommeil, Paris
- Germany (19):
  - Advanced Sleep Research GmbH, Berlin
  - Charite Campus Benjamin Franklin, Klinik und Hochschulambulanz fur Psychiatrie und Psychotherapie, Berlin
  - ClinPharm International GmbH Berlin, Berlin
  - Klinische Forschung Berlin GmbH, Berlin
  - St. Hedwig-Krnkenhaus, Berlin
  - ClinPharm International GmbH Bochum, Bochum
  - ClinPharm International GmbH Chemnitz, Chemnitz
  - ClinPharm International GmbH Dresden, Dresden
  - ClinPharm International GmbH Frankfurt, Frankfurt
  - Department of Psychiatry and Psychotherapy of the University Hospital of Freiburg, Freiburg im Breisgau
  - ClinPharm International GmbH Gorlitz, Görlitz
  - Klinische Forschung, Hamburg
  - ClinPharm International GmbH Leipzig, Leipzig
  - ClinPharm International GmbH Magdeburg, Magdeburg
  - Interdisziplinäres Schlafmedizinisches Zentrum, Universitätsklinikum Giesen und Marburg GmbH, Marburg
  - ClinPharm International GmbH Potsdam, Potsdam
  - Klinik und Poliklinik fur Psychiatre, Regensburg
  - Klinische Forschung Schwerin GmbH, Schwerin
  - SOMNIBENE Institut fur Medizinische, Schwerin
- Hungary (4):
  - Sleep Disorder Centre, State Health Centre, Budapest
  - Department of Neurology , University of Debrecen, Debrecen
  - Dept of Neurology, University of Pecs, Pécs
  - Sleep Laboratory, Ilnd Hospital, Szeged
- Israel (2):
  - Soroka University Medical Center, Unit for Sleep Research, Beersheba
  - Technion Sleep Medicine Center, Rambam Medical Center, Haifa
- Italy (3):
  - IRCCS Neurologico Casimiro Mondino, Centro Multidisciplinare di Medicina del Sonno, Servizio di Neurofisiopatologia, Bologna
  - IRCCS Fondazione San Raffaele del Monte Tabor, Centro per i Disturbi del Sonno, Milan
  - Centro del Sonno, Dipartimento di Neuroscienze, Clinica Neuroligica, Università di Pisa, Pisa
- Poland (6):
  - Klinika Chorob Psychicznych i Zaburzen Nerwicowych ACK, Szpital AMG, Gdansk
  - Laboratorium Diagnostyka Snu, Pro-Medica, Krakow
  - Osrodek Diagnostyki i Leczenia Zaburzen Snu i Chorob Ukladu, Lodz
  - Instytut Psychiatrii i Neurologii, Zaklad Neurofizjologii Klinicznej, Warsaw
  - Laboratorium Diagnostyka Snu, Pro-Medica, Warsaw
  - EMC Instytut Medyczny S.A, Wroclaw
- Slovakia (2):
  - I. Neurologická klinika FNsP Bratislava Nemocnica Staré Mesto, Bratislava
  - Neurologicka klinika, FN L. Pasteura Kosice, Košice
- South Africa (5):
  - BenMed Park Clinic, Benoni, Johannesburg
  - WITS Sleep Laboratory School of Physiology, Parktown, Johannesburg
  - Gatesville Medical Centre, Gatesville, Western Cape
  - Little Company of Mary Hospital, Pretoria
  - Somerset West Trial Centre, Somerset West
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Unidad Framacologia Clinica, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Son Dureta, Unidad de Psicologia, Palma de Mallorca
  - Hospital La Fe, Unidad de Neurofisiologi, Valencia
  - Hospital MAZ, Unidad de Neurofisiologia y Sueno, Zaragoza
- Sweden (3):
  - Carlanderska Sömnlaboratoriet, Gothenburg
  - Örebro University Hospital, Neurology department Sleep Unit, Örebro
  - Aleris Fysiologlab, Stockholm
- Switzerland (5):
  - KSM Zurzach Klinik fur Schlafmedizin, Bad Zurzach
  - Psychiatric University Clinics (UPK) Basel, Sleep Medicine and Neurophysiology, Basel
  - Centre pour l'Etude et le Traitement des Troubles du Sommeil Hopital Bell Idee, Chêne-Bourg
  - KSM Luzern Klinik fur Schlafmedizin, c/o Klinik St. Anna, Lucerne
  - University Hospital Zurich (USZ) Neurology Polyclinic, Center for Sleep Medicine, Zurich
- National Medical University n.a. O.O. BohomoletsChair of Diseases of Nervous System, City Clinical Hospital No.4, Neurological Departments I and II, Kiev, Ukraine
- United Kingdom (2):
  - The Edinburgh Sleep Centre, Edinburgh
  - The London Sleep Centre, London

REFERENCES:
- [Derived] Black J, Pillar G, Hedner J, Polo O, Berkani O, Mangialaio S, Hmissi A, Zammit G, Hajak G. Efficacy and safety of almorexant in adult chronic insomnia: a randomized placebo-controlled trial with an active reference. Sleep Med. 2017 Aug;36:86-94. doi: 10.1016/j.sleep.2017.05.009. Epub 2017 May 29. PMID 28735928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject, first visit was on 28 April 2008. The last subject, last visit (safety follow-up) was on 30 September 2009.
Pre-assignment Details: There was a screening period of 14 to 28 days. Two randomized subjects (one in each almorexant (ACT-078573) dose group) did not receive double-blind study treatment. The 'Started population' was defined as those participants who were randomized and treated.
Groups:
- Placebo: Placebo
  Placebo : 2 placebo matching almorexant tablets and 1 placebo matching over-encapsulated zolpidem
- Almorexant 100mg: almorexant 100 mg
  almorexant : 1 100 mg almorexant tablet, 1 placebo matching almorexant tablet, and 1 placebo matching over-encapsulated zolpidem
- Almorexant 200mg: almorexant 200 mg
  almorexant : 2 100 mg almorexant tablets, and 1 placebo matching over-encapsulated zolpidem
- Zolpidem 10mg: zolpidem 10 mg
  zolpidem : 2 placebo matching almorexant tablets and 1 zolpidem 10 mg over-encapsulated
Period: Overall Study
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Started | 177 (Randomized and started double-blind treatment) | 186 (Randomized and started double-blind treatment) | 176 (Randomized and started double-blind treatment) | 168 (Randomized and started double-blind treatment)
Completed Double-blind Treatment | 163 | 174 | 171 | 161
Completed | 161 (Completed follow-up) | 173 (Completed follow-up) | 170 (Completed follow-up) | 159 (Completed follow-up)
Not Completed | 16 | 13 | 6 | 9
Not completed — Adverse Event | 2 | 7 | 4 | 6
Not completed — Administrative/Other | 7 | 4 | 1 | 2
Not completed — Withdrawal of Consent | 5 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg | Total
Number analyzed (Participants) | 177 | 186 | 176 | 168 | 707
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 177 | 186 | 176 | 168 | 707
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.69) | 44.1 (12.44) | 46.1 (11.83) | 45.1 (12.11) | 45.4 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 113 | 106 | 106 | 436
  Male | 66 | 73 | 70 | 62 | 271
Region of Enrollment [Number; unit: participants]
  Australia | 13 | 15 | 12 | 14 | 54
  Austria | 3 | 5 | 2 | 4 | 14
  Belgium | 0 | 1 | 1 | 0 | 2
  Bulgaria | 1 | 0 | 1 | 0 | 2
  Czech Republic | 2 | 2 | 1 | 1 | 6
  Denmark | 6 | 5 | 5 | 4 | 20
  Finland | 13 | 14 | 13 | 14 | 54
  France | 3 | 2 | 3 | 2 | 10
  Germany | 83 | 86 | 87 | 81 | 337
  Hungary | 12 | 11 | 11 | 13 | 47
  Israel | 5 | 5 | 6 | 5 | 21
  Italy | 3 | 3 | 2 | 2 | 10
  Poland | 3 | 3 | 3 | 3 | 12
  South Africa | 15 | 13 | 13 | 12 | 53
  Spain | 4 | 6 | 5 | 3 | 18
  Sweden | 6 | 8 | 5 | 6 | 25
  Switzerland | 1 | 4 | 4 | 1 | 10
  United Kingdom | 4 | 3 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 1&2 in Wake After Sleep Onset (WASO)
Description: WASO was defined as the time spent in epochs scored as wake after onset of persistent sleep as determined by polysomnography (PSG) until lights on.
  For WASO assessed at the study center, the mean of the 2 PSG nights at each of Visits 3 and 4 was used for Day 1&2 and Day 15&16
Time Frame: From baseline to Day 1&2
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 177 | 186 | 176 | 168
minutes
  Baseline | 85.0 (39.81) [77.3 to 91.0] | 86.6 (39.17) [80.0 to 92.3] | 92.3 (35.92) [84.8 to 98.3] | 76.5 (36.95) [69.3 to 82.0]
  Day 1&2 | 72.8 (42.63) [63.3 to 81.8] | 54.5 (37.65) [47.3 to 61.0] | 46.4 (28.85) [41.8 to 49.8] | 54.6 (36.05) [49.0 to 62.5]
  Change from baseline to day 1&2 | -11.8 (38.73) [-19.3 to -7.3] | -29.0 (31.50) [-33.0 to -23.3] | -40.4 (31.70) [-47.5 to -31.5] | -17.9 (29.19) [-25.3 to -12.0]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -15.0, 95% CI 2-sided [-21.8 to -8.8]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -26.8, 95% CI 2-sided [-34.3 to -19.5]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0376, Wilcoxon rank-sum; Median Difference (Net) = -6.8, 95% CI 2-sided [-13.5 to -0.3]

2. Primary Outcome: Change From Baseline to Day 15&16 in WASO
Description: as for outcome 1
Time Frame: From baseline to Day 15&16
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 177 | 186 | 176 | 168
minutes
  Baseline | 85.0 (39.81) [77.3 to 91.0] | 86.6 (39.17) [80.0 to 92.3] | 92.3 (35.92) [84.8 to 98.3] | 76.5 (36.95) [69.3 to 82.0]
  Day 15&16 | 65.0 (45.90) [56.0 to 71.5] | 55.8 (35.07) [50.5 to 59.0] | 51.8 (31.31) [46.3 to 56.0] | 63.0 (42.31) [56.5 to 72.5]
  Change from baseline to Day 15&16 | -18.3 (43.40) [-22.0 to -12.0] | -29.6 (33.12) [-33.5 to -23.8] | -36.3 (35.20) [-43.8 to -26.5] | -15.1 (36.61) [-19.0 to -8.8]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -13.5, 95% CI 2-sided [-20.3 to -6.5]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -19.5, 95% CI 2-sided [-27.3 to -12.3]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p = 0.3358, Wilcoxon rank-sum; Median Difference (Net) = 3.5, 95% CI 2-sided [-3.8 to 11.0]

3. Primary Outcome: Change From Baseline to Week 1&2 in the Self-reported WASO (sWASO)
Description: sWASO was the self-reported time spent awake after sleep onset as reported in the sleep diary. For sWASO assessed at home, the mean of all available data collected between Visits 3 and 4 (i.e., after the second morning of Visit 3 and before the first evening of Visit 4) was used for Week 1&2
Time Frame: From baseline to Week 1&2
Population: All treated patients with available data
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 175 | 179 | 173 | 168
minutes
  Baseline | 64.0 (51.32) [60.0 to 75.0] | 65.0 (60.49) [59.5 to 72.0] | 69.0 (46.68) [63.0 to 77.0] | 61.6 (48.29) [55.0 to 70.9]
  Week 1&2 | 52.9 (48.33) [47.5 to 58.1] | 40.5 (50.87) [34.5 to 48.3] | 42.9 (42.06) [37.5 to 47.5] | 30.5 (42.26) [25.9 to 39.6]
  Change from baseline to week 1&2 | -14.1 (31.84) [-20.0 to -9.2] | -19.5 (36.93) [-22.9 to -12.7] | -21.8 (32.5) [-28.8 to -17.5] | -23.4 (33.22) [-27.5 to -19.0]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0186, Wilcoxon rank-sum; Median Difference (Net) = -7.3, 95% CI 2-sided [-13.3 to -1.3]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0006, Wilcoxon rank-sum; Median Difference (Net) = -10.4, 95% CI 2-sided [-16.4 to -4.6]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -12.7, 95% CI 2-sided [-18.8 to -6.6]

4. Secondary Outcome: Change From Baseline to Day 1&2 in Latency to Persistent Sleep (LPS)
Description: LPS was defined as the time from the start of the PSG recording to the beginning of the first continuous 20 epochs (i.e., 10 minutes) scored as non-wake (i.e., either sleep stage 1 (S1), sleep stage 2 (S2), slow-wave sleep (SWS), or rapid eye movement sleep(REM)) as determined by PSG
Time Frame: From baseline to Day 1&2
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 177 | 186 | 176 | 168
minutes
  Baseline | 57.3 (41.81) [53.0 to 65.5] | 57.4 (37.03) [52.0 to 63.3] | 54.1 (32.89) [47.5 to 58.3] | 56.5 (34.60) [52.3 to 66.0]
  Day 1&2 | 37.5 (34.64) [32.3 to 44.0] | 28.8 (30.13) [25.0 to 34.5] | 25.0 (21.97) [22.3 to 28.3] | 22.5 (27.25) [20.3 to 26.8]
  Change from baseline to day 1&2 | -15.8 (40.21) [-19.5 to -11.0] | -24.8 (37.00) [-29.8 to -18.3] | -22.5 (30.83) [-27.5 to -20.5] | -29.4 (34.63) [-35.8 to -25.3]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0035, Wilcoxon rank-sum; Median Difference (Net) = -9.3, 95% CI 2-sided [-15.3 to -3.0]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0006, Wilcoxon rank-sum; Median Difference (Net) = -9.5, 95% CI 2-sided [-15.0 to -4.3]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to day 1&2 compared with placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum; Median Difference (Net) = -16.0, 95% CI 2-sided [-22.0 to -9.8]

5. Secondary Outcome: Change From Baseline to Day 15&16 in LPS
Description: as for outcome 4
Time Frame: From baseline to Day 15&16
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 177 | 186 | 176 | 168
minutes
  Baseline | 57.3 (41.81) [53.0 to 65.5] | 57.4 (37.03) [52.0 to 63.3] | 54.1 (32.89) [47.5 to 58.3] | 56.5 (34.60) [52.3 to 66.0]
  Day 15&16 | 30.0 (35.33) [26.0 to 37.8] | 29.3 (28.51) [25.8 to 35.3] | 24.1 (22.48) [21.5 to 28.0] | 24.6 (25.62) [21.3 to 28.3]
  Change from baseline to day 15&16 | -20.0 (46.10) [-25.8 to -16.3] | -23.5 (35.90) [-31.0 to -20.0] | -26.5 (31.10) [-30.8 to -22.8] | -32.3 (34.19) [-36.0 to -26.0]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p = 0.2237, Wilcoxon rank-sum; Median Difference (Net) = -4.0, 95% CI 2-sided [-11.0 to 2.5]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p = 0.0607, Wilcoxon rank-sum; Median Difference (Net) = -6.0, 95% CI 2-sided [-12.3 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to day 15&16 compared with placebo; Test type: Superiority or Other; p = 0.0017, Wilcoxon rank-sum; Median Difference (Net) = -10.5, 95% CI 2-sided [-17.3 to -4.0]

6. Secondary Outcome: Change From Baseline to Week 1&2 in Subjective Latency to Sleep Onset (sLSO)
Description: sLSO was the self-reported time to fall asleep as reported in the sleep diary
Time Frame: From baseline to Week 1&2
Population: All treated patients with available data
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Number analyzed (Participants) | 175 | 179 | 173 | 168
minutes
  Baseline | 58.8 (33.68) [52.0 to 64.5] | 55.0 (50.70) [49.0 to 60.6] | 53.3 (27.93) [50.5 to 58.4] | 50.5 (29.34) [45.2 to 57.0]
  Week 1&2 | 45.0 (31.61) [39.2 to 51.0] | 36.5 (40.64) [32.9 to 41.7] | 34.5 (21.56) [31.5 to 38.3] | 33.3 (21.50) [31.1 to 37.2]
  Change from baseline to week 1&2 | -10.0 (26.89) [-15.1 to -4.7] | -16.2 (34.48) [-19.3 to -12.4] | -16.2 (23.22) [-19.9 to -13.5] | -17.2 (25.67) [-19.9 to -12.3]
Statistical Analysis 1: Comparison: Placebo vs Almorexant 100mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p = 0.1187, Wilcoxon rank-sum; Median Difference (Net) = -4.1, 95% CI 2-sided [-9.1 to 0.9]
Statistical Analysis 2: Comparison: Placebo vs Almorexant 200mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0017, Wilcoxon rank-sum; Median Difference (Net) = -7.1, 95% CI 2-sided [-11.5 to -2.7]
Statistical Analysis 3: Comparison: Placebo vs Zolpidem 10mg; Change from baseline to week 1&2 compared with placebo; Test type: Superiority or Other; p = 0.0121, Wilcoxon rank-sum; Median Difference (Net) = -6.1, 95% CI 2-sided [-10.8 to -1.4]

ADVERSE EVENTS:
Time Frame: All adverse events occurring after the start of study treatment and within 24 hours after the last dose of study treatment
Arm/Group | Placebo | Almorexant 100mg | Almorexant 200mg | Zolpidem 10mg
Serious Adverse Events (participants affected / at risk) | 0/177 | 2/186 | 1/176 | 0/168
Other Adverse Events (participants affected / at risk) | 64/177 | 65/186 | 61/176 | 72/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=177) | Almorexant 100mg (N=186) | Almorexant 200mg (N=176) | Zolpidem 10mg (N=168)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=177) | Almorexant 100mg (N=186) | Almorexant 200mg (N=176) | Zolpidem 10mg (N=168)
HEADACHE (Nervous system disorders) | 21 | 18 | 26 | 29
FATIGUE (General disorders) | 2 | 9 | 6 | 6
DIZZINESS (Nervous system disorders) | 10 | 6 | 8 | 3
SOMNOLENCE (Nervous system disorders) | 4 | 6 | 5 | 4
NAUSEA (Gastrointestinal disorders) | 7 | 4 | 6 | 4
ASTHENIA (General disorders) | 2 | 5 | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 5 | 2 | 5
DIARRHOEA (Gastrointestinal disorders) | 1 | 6 | 1 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 3 | 2 | 1
DEPRESSED MOOD (Psychiatric disorders) | 0 | 2 | 1 | 3
BALANCE DISORDER (Nervous system disorders) | 0 | 1 | 2 | 2
WEIGHT INCREASED (Investigations) | 0 | 0 | 3 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 1 | 3
PARAESTHESIA (Nervous system disorders) | 2 | 1 | 1 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1 | 1 | 2
NIGHTMARE (Psychiatric disorders) | 2 | 0 | 2 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2
PALPITATIONS (Cardiac disorders) | 1 | 1 | 1 | 2
ANXIETY (Psychiatric disorders) | 0 | 1 | 1 | 2
CHEST DISCOMFORT (General disorders) | 1 | 1 | 1 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 1 | 2
BLEPHAROSPASM (Eye disorders) | 0 | 0 | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 0 | 0
FOOD CRAVING (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
INFLUENZA (Infections and infestations) | 0 | 2 | 0 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 1 | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 2 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 1 | 0 | 3
VISION BLURRED (Eye disorders) | 3 | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other